CLINICAL TRIAL: NCT00094211
Title: Neighborhood Impact on Physical Activity in Older Adults
Brief Title: Understanding the Impact of Neighborhood Type on Physical Activity in Older Adults
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Abby C King, Professor, Health Research & Policy and Medicine, Stanford University
Other Study IDs: 1275; R01HL077141 (NIH)
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Low Walkability/Low Income: Participants reside in a low walkability, low income neighborhood
- Low Walkability/High Income: Participants reside in a low walkability, high income neighborhood
- High Walkability/Low Income: Participants reside in a high walkability, low income neighborhood
- High Walkability/High Income: Participants reside in a high walkability, high income neighborhood

SUMMARY:
The purpose of this study is to investigate whether seniors living in neighborhoods that are conducive to walking are more physically active than those living in neighborhoods that are less conducive to walking.

DETAILED DESCRIPTION:
BACKGROUND:

Despite the recognized benefits of regular physical activity for older adults, people over the age of 65 remain among the most inactive groups of the U.S. population. Efforts to understand the factors influencing physical activity in this important group have been limited primarily to demographic and psychosocial domains. The importance of the neighborhood environment in influencing a host of health, behavioral, and psychosocial outcomes has been recognized. However, to date, no systematic investigation of the relationship between objective and subjective environmental factors and objectively measured physical activity levels among older adults has been undertaken.

DESIGN NARRATIVE:

This observational study will investigate whether seniors living in neighborhoods conducive to walking are more physically active, after adjusting for socioeconomic status (SES), than those living in neighborhoods less conducive to walking or other forms of physical activity for transportation or recreational purposes. Additional questions of interest concern the moderating effects of physical function and the proportion of seniors living nearby on the relationship between environment and physical activity. The study will take advantage of the sampling, recruitment, and data collection methods of an ongoing NIH-funded research project aimed at integrating public health and urban planning frameworks in studying the impacts of environmental factors on physical activity levels in younger adults. Population-based sampling methods will be used to recruit adults over 65 years of age who are living in more walkable versus less walkable neighborhoods of varying SES levels. Participants will be recruited from Seattle, Washington (n = 600) and Baltimore, Maryland (n = 600). In addition to objectively measured physical environment (using geographic information systems {GIS}) and physical activity levels (using accelerometry), self-reported neighborhood environment, physical activity, and quality of life variables of particular relevance to older adults will be assessed twice during a 12-month period.

ELIGIBILITY:
Inclusion criteria:

* Currently living in an apartment, condo, house, or assisted living facility
* Able to walk more than 10 feet at a time
* Able to speak and read English
* Able to complete study surveys (with assistance if necessary)

Exclusion Criteria:

* Not currently living in one of the areas in which the study will take place

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Residents of selected block groups in King County, WA and the Baltimore region.
Sampling Method: Non-Probability Sample
Enrollment: 896 (Actual)
Dates: Start 2004-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby King, Principal Investigator — Stanford University
Locations (3):
- United States (2):
  - San Diego State University, San Diego, California
  - Stanford University School of Medicine, Stanford, California
- University of British Columbia-Vancouver, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Stewart AL, Mills KM, King AC, Haskell WL, Gillis D, Ritter PL. CHAMPS physical activity questionnaire for older adults: outcomes for interventions. Med Sci Sports Exerc. 2001 Jul;33(7):1126-41. doi: 10.1097/00005768-200107000-00010. PMID 11445760

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 896 participants were enrolled in the the study, but 34 dropped out after receiving the study materials and before completing the measures. Therefore, 862 participants provided data for this study.
Groups:
- High Walkability/High Income: Households were enumerated in King County, WA and in the Baltimore, MD-Washington, DC area based on geographical information systems-derived walkability index and neighborhood-level income. Four quadrants were derived based on these two factors: higher walkability-higher income; higher walkability-lower income; lower walkability-higher income; and lower walkability-lower income neighborhoods. This arm represents the High Walkability/High Income quadrant.
- High Walkability/Low Income; Low Walkability/Low Income: Households were enumerated in King County, WA and in the Baltimore, MD-Washington, DC area based on geographical information systems-derived walkability index and neighborhood-level income. Four quadrants were derived based on these two factors: higher walkability-higher income; higher walkability-lower income; lower walkability-higher income; and lower walkability-lower income neighborhoods. This arm represents the High Walkability/Low Income quadrant.
- Low Walkability/High Income: Households were enumerated in King County, WA and in the Baltimore, MD-Washington, DC area based on geographical information systems-derived walkability index and neighborhood-level income. Four quadrants were derived based on these two factors: higher walkability-higher income; higher walkability-lower income; lower walkability-higher income; and lower walkability-lower income neighborhoods. This arm represents the Low Walkability/High Income quadrant.
Period: Overall Study
Arm/Group | High Walkability/High Income | High Walkability/Low Income | Low Walkability/High Income | Low Walkability/Low Income
Started | 221 | 259 | 230 | 186
Completed | 212 | 251 | 220 | 179
Not Completed | 9 | 8 | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- High Walkability/High Income; High Walkability/Low Income; Low Walkability/High Income; Low Walkability/Low Income: Households were enumerated in King County, WA and in the Baltimore, MD-Washington, DC area based on geographical information systems-derived walkability index and neighborhood-level income. Four quadrants were derived based on these two factors: higher walkability-higher income; higher walkability-lower income; lower walkability-higher income; and lower walkability-lower income neighborhoods.
- Total: Total of all reporting groups
Arm/Group | High Walkability/High Income | High Walkability/Low Income | Low Walkability/High Income | Low Walkability/Low Income | Total
Number analyzed (Participants) | 212 | 251 | 220 | 179 | 862
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 212 | 251 | 220 | 179 | 862
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (7.1) | 75.7 (6.8) | 74.6 (6.8) | 75.0 (6.5) | 75.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 155 | 109 | 103 | 482
  Male | 97 | 96 | 111 | 76 | 380
Region of Enrollment [Number; unit: participants]
  United States | 212 | 251 | 220 | 179 | 862

OUTCOME MEASURES:

1. Primary Outcome: Physical Environment Factors Using Geographic Information Systems [GIS]
Description: Physical environment factors measured using GIS-derived measures of street connectivity, residential density, and mixed land use in participant block groups and a network buffer around each participant's home. A walkability index was created for a 500 meter street network buffer around participant homes. The walkability index was calculated for each census block group in the regions by summing the z-scores of four macro built environment measures: 1) net residential density, 2) intersection density, 3) retail floor to land area ratio (FAR), and 4) mixed use. A higher scores indicates higher walkability. The minimum value is -4.08 and the maximum value is 12.5.
Time Frame: at two time points, 6 months apart, which were averaged
Population: GIS variables were created for all participants enrolled in the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Walkability/High Income | High Walkability/Low Income | Low Walkability/High Income | Low Walkability/Low Income
Number analyzed (Participants) | 221 | 259 | 230 | 186
units on a scale | 1.3 (3.0) | 1.9 (3.2) | -2.1 (1.0) | -1.6 (1.2)

2. Primary Outcome: Community Healthy Activities Model Program for Seniors (CHAMPS) Self-reported Walking for Errands
Description: A self-report physical activity questionnaire that assesses weekly frequency and duration of various activities typically undertaken by midlife and older adults over the prior 4-week period. Self-reported walking for errands is one physical activity item assessed. The measure has been shown to have good test-retest reliability (stability) and construct and concurrent validity, and has been shown to be sensitive to change in a variety of adult populations. It has seven frequency categories (from less than 1 hour a week to 9 or more hours per week). The minimum value is 0 and the maximal value is variable. (See Stewart AL, Mills KM, King AC, et al. CHAMPS Physical Activity Questionnaire for Older Adults: Outcomes for Interventions. Med Sci Sports Exerc, 33:7, 1126-1141, 2001.)
Time Frame: Assessment at baseline and 6 months, with the data across these two time points averaged to increase outcome stability.
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | High Walkability/High Income | High Walkability/Low Income | Low Walkability/High Income | Low Walkability/Low Income
Number analyzed (Participants) | 216 | 257 | 228 | 182
minutes per week | 80.6 (106.7) | 46.3 (84.3) | 21.5 (55.8) | 21.5 (66.2)

3. Primary Outcome: Accelerometer Measured Physical Activity
Description: Ambulatory assessment of moderate-to-vigorous physical activity using a validated Actigraph accelerometer. Participants were instructed to wear the accelerometer during waking hours for seven days at each of the two measurement points. The accelerometer was placed over the right hip. Data were cleaned and scored using MeterPlus version 4.0 software.
Time Frame: Assessment at baseline and 6 months, with the data across these two time points averaged to increase outcome stability.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | High Walkability/High Income | High Walkability/Low Income | Low Walkability/High Income | Low Walkability/Low Income
Number analyzed (Participants) | 212 | 251 | 220 | 179
minutes per day | 17.2 (18.5) | 8.9 (12.6) | 13.5 (15.7) | 10.3 (15.6)

4. Primary Outcome: Neighborhood Environment for Walkability Survey (NEWS) - Walking and Cycling Facilities in Neighborhood
Description: The scale is walking/cycling facilities which is a mean of 5 items. The minimum value is 1 and the maximum value is 4. Higher scores indicate an environment that is supportive of walking and cycling which is a better outcome.
Time Frame: Assessment at baseline and 6 months, with the data across these two time points averaged to increase outcome stability.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Walkability/High Income | High Walkability/Low Income | Low Walkability/High Income | Low Walkability/Low Income
Number analyzed (Participants) | 212 | 250 | 220 | 179
units on a scale | 3.2 (0.6) | 2.9 (0.7) | 2.6 (0.9) | 2.4 (0.9)

5. Primary Outcome: Neighborhood Environment for Walkability Survey (NEWS) - Land Use Mix Access
Description: The scale is land use mix access which is a mean of 7 items. The minimum value is 1 and the maximum value is 4. Higher scores indicate easier access to services which is indicative of a high walkability environment (i.e., a better outcome).
Time Frame: Assessment at baseline and 6 months, with the data across these two time points averaged to increase outcome stability.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Walkability/High Income | High Walkability/Low Income | Low Walkability/High Income | Low Walkability/Low Income
Number analyzed (Participants) | 212 | 251 | 220 | 179
units on a scale | 3.1 (0.5) | 2.9 (0.5) | 2.4 (0.6) | 2.5 (0.6)

ADVERSE EVENTS:
Time Frame: 2 years, 9 months
Groups:
- High Walkability/High Income; High Walkability/Low Income; Low Walkability/High Income; Low Walkability/Low Income: Households were enumerated in King County, WA and in the Baltimore, MD-Washington, DC area based on geographical information systems-derived walkability index and neighborhood-level income. Four quadrants were derived based on these two factors: higher walkability-higher income; higher walkability-lower income; lower walkability-higher income; and lower walkability-lower income neighborhoods.
  There were no treatment conditions in this cross-sectional observational study. No adverse events were reported.
Arm/Group | High Walkability/High Income | High Walkability/Low Income | Low Walkability/High Income | Low Walkability/Low Income
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/251 | 0/220 | 0/179
Other Adverse Events (participants affected / at risk) | 0/212 | 0/251 | 0/220 | 0/179

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No